CLINICAL TRIAL: NCT01031654
Title: Marital Functioning Among Combat Veterans
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cheryl Gore-Felton, Professor, Stanford University
Other Study IDs: SU-04222009-2379; 9022 (Other: Stanford University IRB)
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of this research study is to examine marital dynamics related to husband-wife reunification following the veteran's return

DETAILED DESCRIPTION:
We are interested in patterns of husband/wife communication and interaction regarding conflict resolution, trauma experiences, marital satisfaction, occupational functioning, social functioning, family functioning, and substance use.

We hope to discover ways to assist couples in reducing marital stress.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Married or in a married like relationship
* One partner has served in Afghanistan or Iraq

Exclusion Criteria:

* Separated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 10 couples (N=20) will be enrolled in the study. At least one of the marital dyad will be an Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) veteran.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Gore-Felton Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States